CLINICAL TRIAL: NCT01124903
Title: Human Hydration Status Monitoring: Phase I
Brief Title: Human Hydration Status Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: ChromoLogic, LLC (Industry); Intelligent Automation, Inc. (Industry); Gaia Medical Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H08-12
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Dehydration
Keywords: dehydration; hypohydration; diagnostic accuracy; biological variation; hydration assessment; body mass; osmolality; plasma; saliva; urine
MeSH Terms: conditions — Dehydration | interventions — Organism Hydration Status

STUDY DESIGN:
Intervention Model Description: single-sample pre-post design
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dehydration (Experimental): Multiple measures of hydration status were made when subjects were normally hydrated (euhydrated) and when dehydrated. The diagnostic usefulness of the measures was determined.
  Interventions: Procedure: Dehydration

INTERVENTIONS:
Procedure: Dehydration — Subjects were dehydrated by 2 - 7% of body mass over 3-5 hours using exercise-heat stress and fluid restriction.
  Other Names: Hypohydration

SUMMARY:
The sports medicine literature provides a consensus on what threshold values constitute euhydration (normal body water) using a variety of hydration assessment markers (e.g., blood, urine). The investigators add to this literature by providing decision levels for multiple body fluids which can be used as starting points for diagnosing and treating dehydration. At present, plasma osmolality (Posm) provides the best potential measure for static dehydration assessment (spot measure), while dynamic dehydration assessment (serial monitoring) is best accomplished using change values for Posm, urine specific gravity, or body mass (weight). These findings should be considered useful for clinical, military, and sports medicine communities.

DETAILED DESCRIPTION:
Well-recognized markers for static (one time) or dynamic (monitoring over time) dehydration assessment have not been rigorously tested for their usefulness in clinical, military, and sports medicine communities.

This study evaluated the components of biological variation and accuracy of potential markers in plasma, urine, saliva, and body mass, for static and dynamic dehydration assessment. Design: Eighteen healthy volunteers (13M, 5F) were studied while carefully controlling hydration and numerous pre-analytical factors. Biological variation was determined over three consecutive days using published methods. Atypical values based on statistical deviations from a homeostatic set-point were examined. Measured deviations in body fluid were produced using a separate, prospective dehydration experiment and evaluated by ROC analysis to quantify diagnostic accuracy.

All dehydration markers displayed substantial individuality and half displayed marked heterogeneity of intra-individual variation. Decision levels for all dehydration markers were within one standard deviation of the ROC criterion values and most were nearly identical to the prospective group means after dehydrating volunteers by 1.8 - 7.0% of body mass. However, only plasma osmolality (Posm) showed statistical promise for use in static dehydration assessment. A 301 ± 5 mmol/kg diagnostic decision level is proposed. Reference change values (RCV) of 9 mmol/kg (Posm), 0.010 (urine specific gravity, Usg), and 2.5% change in body mass (Bm) were also statistically valid for dynamic dehydration assessment at the 95% probability level.

Posm is the only useful marker for static dehydration assessment. Posm, Usg, and Bm are valid markers in the setting of dynamic dehydration assessment.

ELIGIBILITY:
Inclusion Criteria:

* You are a member of the U.S. Army between 18-39 years of age
* You have passed the APFT within the previous 12 months
* You have completed and passed a recent medical physical exam
* You are willing to discuss with OMSO and the Principle Investigator (PI) all medications and supplements you are taking and you are willing to stop taking any supplements not approved by OMSO and the PI.

Exclusion Criteria:

* You have any physical problems that would make exercise difficult
* You have ever had a heat injury or have a history of having trouble in the heat
* You have an allergy to sulfa drugs
* You have been treated for dry eyes
* You are pregnant, planning on becoming pregnant during the study, or are presently lactating

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evidence of clinical dehydration | 24 hours
  Dehydration was carefully imposed in healthy human subjects. The diagnostic usefulness of multiple classic and novel dehydration assessment measures was made.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Cheuvront, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States